CLINICAL TRIAL: NCT06067230
Title: A Phase 3 Study to Evaluate the Immunogenicity and Safety of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus, in High-Risk Adults
Brief Title: A Study to Investigate the Immunogenicity and Safety of mRNA-1345 Vaccine Targeting Respiratory Syncytial Virus (RSV) in High-risk Adults
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P303
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Respiratory syncytial virus; Safety; Vaccines; Immunocompromised; Organ transplant
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Intervention Model Description: Part A participants will be randomized into 2 treatment dose groups at a 1:1 ratio.
  Part B is non-randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A: double-blind Part B: open-label (no masking)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: mRNA-1345 Dose 1 (Experimental): Single injection of mRNA-1345 administered intramuscularly (IM) on Day 1.
  Interventions: Biological: mRNA-1345
- Part A: mRNA-1345 Dose 2 (Experimental): Single injection of mRNA-1345 administered IM on Day 1.
  Interventions: Biological: mRNA-1345
- Part B: mRNA-1345 Dose 2 (Experimental): Two injections of mRNA-1345 administered IM on Day 1 and Day 57.
  Interventions: Biological: mRNA-1345

INTERVENTIONS:
Biological: mRNA-1345 — Sterile liquid for injection

SUMMARY:
The study is divided into 2 parts (Part A and Part B). Part A of the study will evaluate the safety and immune response to mRNA-1345 in high-risk adults aged ≥18 to <60 years.

Part B of the study will evaluate the safety and immune response to mRNA-1345 in adults who received solid organ transplant (SOT).

ELIGIBILITY:
Key Inclusion Criteria:

Part A:

* Adults ≥18 to <60 years of age at the time of consent who are primarily responsible for self-care and activities of daily living.
* Documented confirmation by a physician of the diagnosis of at least one of the following conditions:

  1. Coronary artery disease and/or congestive heart failure.
  2. Chronic lung disease (for example, including but not limited to chronic obstructive pulmonary disease or persistent asthma).
  3. Stable type 1 or type 2 diabetes mellitus controlled with at least 1 medication started 90 days or more prior to Day 1.

Part B:

* Adults ≥18 years of age at the time of consent who are primarily responsible for self-care and activities of daily living.
* Recipient of an SOT (kidney, liver, or lung transplant) ≥180 days prior to day of consent and receiving chronic immunosuppressive therapy for the prevention of allograft rejection.

Parts A and B:

- Able to comply with study requirements.

Key Exclusion Criteria:

Part A:

* Participation in an another clinical research trial where the participant has received an investigational product 180 days prior to Day 1. Participation in an RSV trial at any time prior to Day 1 is exclusionary.
* History of a diagnosis or condition, that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of the mRNA-1345 injection or any components of the mRNA-1345 injection.
* Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 180 days prior to Day 1.
* History of myocarditis, pericarditis, or myopericarditis.

Part B:

* Previous treatment with alemtuzumab or rituximab within 2 years prior to Day 1.
* Previous treatment with plasmapheresis within 30 days prior to Day 1.
* A history of complications of immunosuppression.
* A history of biopsy proven or clinically diagnosed rejection within 90 days prior to Day 1 or suspected active chronic rejection according to the Investigator's judgment.

Note: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Day 1 through Day 7 (7 days post injection) for Part A and Day 1 through Day 64 (7 days post second injection) for Part B
Number of Participants with Unsolicited Adverse Events (AEs) | Day 1 through Day 28 (28 days post injection) for Part A and Day 1 through Day 84 (28 days post second injection) for Part B
Number of Participants With Medically Attended AEs (MAAEs) | Day 1 through Month 6 (for Part A) and Day 1 through Month 9 (for Part B)
Number of Participants With Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), and AEs Leading to Discontinuation | Day 1 through End of Study (Day 730)
Part A: Geometric Mean Titer (GMT) of Serum Respiratory Syncytial Virus Subtype A (RSV-A) and Respiratory Syncytial Virus Subtype B (RSV-B) Neutralizing Antibodies (Abs) at Day 29 | Day 29
Part B: GMT of Serum RSV-A and RSV-B Neutralizing Abs at Day 85 | Day 85

SECONDARY OUTCOMES:
Part A: Seroresponse Rate (SRR) of RSV-A and RSV-B Neutralizing Abs on Day 29 | Day 29
Part A: Geometric Mean Concentration (GMC) of Serum RSV Prefusion Conformation of the F Protein (Pre-F) Binding Abs | Up to End of Study (Day 730)
Part A: Geometric Mean Fold-Rise (GMFR) of Serum RSV Pre-F Binding Abs | Up to End of Study (Day 730)
Part A: SRR of Serum RSV Pre-F Binding Abs at Postbaseline/Baseline Levels | Baseline up to Day 730
Part A: Number of Participants with ≥2-Fold Increase in RSV Pre-F Binding Abs | Up to End of Study (Day 730)
Part A: GMT of Serum RSV-A and RSV-B Neutralizing Abs at Day 29 | Day 29
Part A: GMT of Postinjection/Baseline Titers to RSV-A and RSV-B Neutralizing Abs | Baseline up to Day 730
Part A: GMFR of Postinjection/Baseline Titers to RSV-A and RSV-B Neutralizing Abs | Baseline up to Day 730
Part A: SRR of Serum RSV-A and RSV-B Neutralizing Abs | Up to End of Study (Day 730)
Part A: Number of Participants with ≥2-Fold Increase in RSV-A and RSV-B Neutralizing Abs Titers | Up to End of Study (Day 730)
Part B: GMT of Serum RSV-A and RSV-B Neutralizing Abs at Day 29 | Day 29
Part B: SRR of Serum RSV-A and RSV-B Neutralizing Abs on Day 29 | Day 29
Part B: SRR of Serum RSV-A and RSV-B Neutralizing Abs on Day 85 | Day 85
Part B: GMT of Serum RSV-A and RSV-B Neutralizing Abs | Up to End of Study (Day 730)
Part B: GMFR of Serum RSV-A and RSV-B Neutralizing Abs | Up to End of Study (Day 730)
Part B: SRR of Serum RSV-A and RSV-B Neutralizing Abs at Postbaseline/Baseline Levels | Baseline up to Day 730
Part B: Number of Participants with ≥2-Fold Increase in RSV-A and RSV-B Neutralizing Abs | Up to End of Study (Day 730)
Part B: GMC of Serum RSV Pre-F Binding Abs | Up to End of Study (Day 730)
Part B: GMFR of Serum RSV Pre-F Binding Abs | Up to End of Study (Day 730)
Part B: SRR of Serum RSV Pre-F Binding Abs at Postbaseline/Baseline Levels | Baseline up to End of Study (Day 730)
Part B: Number of Participants with ≥2-Fold Increase in RSV Pre-F Binding Abs | Up to End of Study (Day 730)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (32):
  - Lenzmeier Family Medicine - CCT - PPDS, Glendale, Arizona
  - Foothills Research Center - CCT - PPDS, Phoenix, Arizona
  - Fiel Family & Sports Medicine - PC - CCT - PPDS, Tempe, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Artemis Institute For Clinical Research LLC - San Diego - Headlands - PPDS, San Diego, California
  - Critical Care, Pulmonary and Sleep Associates / CCT Research, Lakewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Excel Medical Clinical Trials DBA Flourish, Boca Raton, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - CenExel RCA - Hollywood, Hollywood, Florida
  - Clinical Research Atlanta - Headlands - PPDS, Stockbridge, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - University of Chicago, Chicago, Illinois
  - AES - DRS - Optimal Research Illinois - Peoria, Peoria, Illinois
  - Benchmark Research - Covington - HyperCore - PPDS, Covington, Louisiana
  - Velocity Clinical Research (Rockville - Maryland) - PPDS, Rockville, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - DM Clinical Research - Southfield - ERN - PPDS, Southfield, Michigan
  - Velocity Clinical Research (Lincoln - Nebraska) - PPDS, Lincoln, Nebraska
  - University of Rochester - Rochester General Hospital - PPDS, Rochester, New York
  - Montefiore Medical Center - BRANY - PPDS, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - DM Clinical Research - Philadelphia - ERN - PPDS, Philadelphia, Pennsylvania
  - Benchmark Research - Fort Worth - HyperCore - PPDS, Fort Worth, Texas
  - DM Clinical Research - Cyfair Clinical Research Center, Houston, Texas
  - Benchmark Research - San Angelo - HyperCore - PPDS, San Angelo, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - Springville Dermatology - CCT - PPDS, Springville, Utah
  - Velocity Clinical Research - Hampton - PPDS, Hampton, Virginia
  - Centricity Research Suffolk Family Medicine, Suffolk, Virginia
  - Velocity Clinical Research - Family Practice - Suffolk - PPDS, Suffolk, Virginia
- Canada (6):
  - University of Alberta, Edmonton, Alberta
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Colchester Research Group, Truro, Nova Scotia
  - Diex Recherche - Sherbrooke - PPDS, Sherbrooke, Quebec
  - Diex Recherche - Québec - PPDS, Québec
- Caribbean Medical Research Center, San Juan, Puerto Rico
- United Kingdom (5):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Fylde Coast Clinical Research, Blackpool, Lancashire
  - Liverpool School of Tropical Medicine, Liverpool, Merseyside
  - Aberdeen Royal Infirmary - PPDS, Aberdeen
  - The Royal Free Hospital, London

REFERENCES:
- [Derived] Mayer EF, Falsey AR, Clark R, Ferguson M, Cardona J, She F, Jones B, Reuter C, Collins A, Mannan A, Kapoor A, Slobod K, Stoszek SK, Du J, Mou J, Lan L, Zhou H, Wilson E, Goswami J, Das R, Priddy F. Safety, Tolerability, and Immunogenicity of mRNA-1345 in Adults at Increased Risk for RSV Disease Aged 18 to 59 Years. Clin Infect Dis. 2025 Jun 4:ciaf292. doi: 10.1093/cid/ciaf292. Online ahead of print. PMID 40464662